CLINICAL TRIAL: NCT06905431
Title: Effects of Plyometric and High Intensity Interval Training on Sprint Speed, Agility and Power Among Female Fast Bowlers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/784
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Health Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior | interventions — Plyometric Exercise; High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric Training (Experimental)
  Interventions: Diagnostic Test: Plyometric Training
- High-Intensity Interval Training (HIIT) (Active Comparator)
  Interventions: Combination Product: (High-Intensity Interval Training (HIIT)

INTERVENTIONS:
Diagnostic Test: Plyometric Training — Frequency: Three sessions per week on non-consecutive days to allow for adequate recovery.
  Intensity: High-intensity exercises performed at 80-90% of maximum effort. Exercises include box jumps, depth jumps, lateral bounds, and tuck jumps targeting explosive power and agility.
  Time: Each session lasts approximately 45-60 minutes, including: Warm-up (10 minutes), Core Plyometric Exercises (30-40 minutes), Cool-down (5-10 minutes) Type: Explosive lower-body movements utilizing the stretch-shortening cycle (SSC) to improve neuromuscular coordination, sprint speed, and power."
  Arms: Plyometric Training
Combination Product: (High-Intensity Interval Training (HIIT) — Frequency: Three sessions per week (e.g., Tuesday, Thursday, Saturday) with a rest day between sessions. Intensity: Alternating between 85-95% of maximum heart rate during high-intensity intervals and 50-60% of maximum heart rate during recovery periods. Work-to-rest ratio of 1:2 (e.g., 30 seconds of high-intensity sprints followed by 60 seconds of low-intensity walking). Time: Each session lasts approximately 45-50 minutes, including: Warm-up (10 minutes), HIIT Intervals (25-30 minutes with 8-12 work-rest cycles), Cool-down (5-10 minutes) Type: Cardiovascular exercises such as sprinting, cycling, or shuttle runs designed to enhance anaerobic capacity, agility, and sprint speed.
  Arms: High-Intensity Interval Training (HIIT)

SUMMARY:
This study will investigate the comparative effects of plyometric training (PT) and high-intensity interval training (HIIT) on key performance metrics: sprint speed, agility, and power. The research will be conducted as a randomized clinical trial over six months, involving 34 participants recruited from cricket academies.

DETAILED DESCRIPTION:
Participants will be randomly assigned to either the PT or HIIT group. The PT group will perform exercises leveraging the stretch-shortening cycle to enhance explosive power, while the HIIT group will alternate high-intensity activity with recovery periods to improve anaerobic capacity. Standardized tools, including the 40-Yard Sprint Test, Standing Broad Jump, and Agility T-Test, will be used to assess outcomes pre- and post-intervention. Data will be analyzed using SPSS, employing paired t-tests and Mann-Whitney U tests for within- and between-group comparisons

ELIGIBILITY:
Inclusion Criteria:

* Female fast bowlers age 18-25 years
* Active cricketers with at least 2 years of experience in fast bowling (20)
* Active health status, no history of severe injuries

Exclusion Criteria:

* Any history of chronic injuries, musculoskeletal disorders, or conditions that could be exacerbated by high-intensity exercise.
* Participants not regularly training or competing in cricket.
* Females underwent C-section and or having two children will exclude

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
40 Yard Sprint Test | 12 Months
  The 40-Yard Sprint Test is a reliable and valid assessment to measure an individual's speed and acceleration over a 40-yard distance, commonly used in sports like football and cricket. Participants sprint maximally from a stationary start, with the time recorded using a stopwatch or timing gates. The best time from 2-3 trials is used for scoring, with elite athletes completing the test in approximately 4.5-5.5 seconds. Highly reliable when standardized conditions are applied, the test provides valuable insights into an athlete's speed capabilities, making it a critical tool for performance evaluation and training program effectiveness.
Standing Broad Jump (SBJ) | 12 Months
  The Standing Broad Jump (SBJ) is a simple yet effective test to measure explosive lower-body power, widely used in sports and fitness assessments. Participants jump forward as far as possible from a stationary position, using arm swings and leg power, with the distance measured from the starting line to the nearest point of contact on landing. Typically performed in 2-3 attempts, the best score is recorded. The SBJ is highly reliable under standardized conditions and valid for evaluating leg strength and performance in sports requiring explosive movements. It is a valuable tool for tracking progress in athletic training and rehabilitation.
Assessment of Agility T-Test | 12 Months
  The Agility T-Test is a widely used fitness assessment to measure agility, focusing on an individual's ability to change direction quickly while maintaining control. It involves sprinting, lateral shuffles, and backpedaling between four cones arranged in a ""T"" shape. Participants start at the base cone, sprint forward, shuffle laterally to the left and right cones, return to the central cone, and backpedal to the starting point. The test is scored based on time, with faster times indicating better agility. Highly reliable and valid, the T-Test is commonly used to assess and improve multidirectional movement skills in sports and fitness programs

CONTACTS AND LOCATIONS:
Locations (1):
- Punjab university, education university, GCU university, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No